CLINICAL TRIAL: NCT00476528
Title: Early Rehabilitation of Patients With Posttraumatic Amnesia. A Clinical Controlled Investigation of the Effect of a Nursing Programme in Patients With Traumatic Brain Injury in the Acute Care
Brief Title: Early Rehabilitation of Patients With Posttraumatic Amnesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Jens Christian Sorensen, Professor, Aarhus University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NK8633
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Amnesia
Keywords: Posttraumatic amnesia; Early intervention; A systematic nursing programme in the ICU; Early identification of patients with posttraumatic amnesia
MeSH Terms: conditions — Amnesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Reality Orientation — Two matched groups of patients diagnosed with TBI are selected from two university hospitals. In addition to conventional treatment, patients in one group are introduced to a reality- orientation programme consisting of systematic orientation, information, and systematic cooperation with the patient´s relatives.Patients in the other group receive conventional treatment only. All patients are tested on a daily basis in accordance with the RLAS and the GOAT test.
Behavioral: Reality Orientation — A quasiexperimental study

SUMMARY:
The purpose of this study is to investigate if a systematic intervention with early identifying of patients with posttraumatic amnesia using a reality orientation therapy can reduce the period with posttraumatic amnesia in order to get a better outcome for patients with traumatic brain injury

DETAILED DESCRIPTION:
1. A systematic review with the latest investigation and treatment of patients with posttraumatic amnesia
2. Investigate the effect of a systematic nursing programme on the length of posttraumatic amnesia
3. Investigate the effect of a systematic nursing programme after 12 month
4. Describe perspectives for the future within the early rehabilitation of patients with posttraumatic amnesia

ELIGIBILITY:
Inclusion Criteria:

* Patients should be able to speak and understand danish
* Patients with traumatic brain injury
* A verified brain injury at the CT scanning

Exclusion Criteria:

* Patients with medical illness
* Patients with other neurological illness
* Patients with neuroinfections meningitic, encephalitic
* Patients who does not understand and speaks danish

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Duration of posttraumatic amnesia Results of score with RLAS, GOAT, GOSE and LOS | 12month

CONTACTS AND LOCATIONS:
Overall Officials: Jens Christian Soerensen, Study Director — Department of Neurosurgery NK
Locations (1):
- University Hospital, Aarhus, Central Jutland, Denmark